CLINICAL TRIAL: NCT05551338
Title: Serious Games for Parkinson's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Jean-Francois Daneault, Ph.D., Assistant professor, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro2020002765
Record Dates: First submitted 2022-06-21; First posted 2022-09-22 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-09

CONDITIONS: Parkinson Disease; Parkinson
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: Group 1: 10 patients will be asked to perform two 30-minute sessions per week of training using serious games over a 3-month period in addition to their conventional care.
  Group 2: 10 patients will only receive their conventional care.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors will be blinded to participant assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Patients will be asked to perform two 30-minute sessions per week of training using serious games over a 3-month period in their home setting in addition to their conventional care
  Interventions: Other: Serious games
- Control (No Intervention): Patients will undergo only their conventional care

INTERVENTIONS:
Other: Serious games — The training protocol will entail using a tablet-based program that includes 6 serious games. Patients will be asked to use the program twice a week for 3 months. The serious games that will be used in this study were developed to challenge short-term memory and selective attention in six different games. Each of the six games comprise 20 different stages of varying difficulty, where stage 1 is the easiest and stage 20 is the most difficult.
  Arms: Intervention

SUMMARY:
IMPORTANCE: Rehabilitation games have been shown to improve cognitive function among people with various disorders but they have not been explored in home settings for patients with Parkinson's disease.

OBJECTIVE: To collect pilot data regarding the therapeutic benefits of self-administered rehabilitation games among patients with Parkinson's disease.

METHODS: The investigators will recruit 20 patients with Parkinson's disease into a pilot randomized controlled trial. Patients will be asked to perform two 30-minute sessions per week of training using serious games over a 3-month period in addition to conventional care or undergo only usual care. Patients will be evaluated at baseline, after 12 weeks of treatment, and at 24 weeks. Improvements in cognitive function, depression, quality of life, and mobility will be assessed.

RELEVANCE: Identifying whether self-administered rehabilitation games can lead to clinical improvements could have significant implications for the management of the disease.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of mild to moderate PD (Hoehn & Yahr 1-3)
2. baseline MoCA score <26
3. ≥ 18 years-old
4. ability to communicate and read in English
5. have self-reported technological literacy (ie answer yes to the question asking if they are comfortable using technological devices)

Exclusion Criteria:

1. comorbid conditions that could affect the performance of the tasks (e.g. severe uncorrected vision impairment)
2. severe cognitive impairment that would prevent the patient from understanding the tasks (MoCA<16)
3. if the subject does not want to be video recorded during the assessments or interview sessions
4. if the subject does not have access to WiFi

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-06-15 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Montreal Cognitive Assessment (MoCA) | Baseline (week 0)
  The Montreal Cognitive Assessment is a widely used test of cognitive function among the elderly; it includes tests of orientation, attention, memory, language and visual-spatial skills. The minimum score is 0 the maximum score is 30. Higher scores indicate higher cognitive function and lower scores indicate lower cognitive function.
Montreal Cognitive Assessment (MoCA) | Post-intervention (week 12)
  The Montreal Cognitive Assessment is a widely used test of cognitive function among the elderly; it includes tests of orientation, attention, memory, language and visual-spatial skills. The minimum score is 0 the maximum score is 30. Higher scores indicate higher cognitive function and lower scores indicate lower cognitive function.
Montreal Cognitive Assessment (MoCA) | Follow-up (week 24)
  The Montreal Cognitive Assessment is a widely used test of cognitive function among the elderly; it includes tests of orientation, attention, memory, language and visual-spatial skills. The minimum score is 0 the maximum score is 30. Higher scores indicate higher cognitive function and lower scores indicate lower cognitive function.

SECONDARY OUTCOMES:
Digit span forward and backward | Baseline (week 0), Post-intervention (week 12), Follow-up (week 24)
  These tests are used to measure working memory's number storage capacity.
Semantic fluency test | Baseline (week 0), Post-intervention (week 12), Follow-up (week 24)
  This verbal fluency test has been shown to be effective in measuring executive functioning and language ability because the semantic/category subtest seems to require a higher level of thought processes since people have to think of meaning.
Geriatric depression scale | Baseline (week 0), Post-intervention (week 12), Follow-up (week 24)
  The geriatric depression scale is a self-report measure of depression in older adults. The minimum score is 0 and the maximum score is 15. Higher scores indicate greater severity of depressive symptoms and lower scores indicate lesser severity of depressive symptoms.
LifeSpace Assessment | Baseline (week 0), Post-intervention (week 12), Follow-up (week 24)
  The LifeSpace Assessment assesses mobility from the spaces that older adults go, and how often, and how independently they move. The minimum score is 0 and the maximum score is 120. Higher scores indicate a larger life space and lower scores indicate a smaller life space.
PDQ-39 | Baseline (week 0), Post-intervention (week 12), Follow-up (week 24)
  It is a self-administered questionnaire to assess PD-specific health-related quality of life. The 39-item self-report questionnaire will be used to asses quality of life. The questionnaire has 8 domains (e.g. mobility, emotional well-being, stigma, social support, cognition, communication, and bodily discomfort). It contains questions asking how often certain difficulties/problems have occurred within the last month with answers ranging from "never" to "always." Each dimension total score ranges from 0 (never have difficulty) to 100 (always have difficulty). Higher scores indicate poorer quality of life and lower scores indicate higher quality of life.
Sensor-based mobility | Baseline (week 0), Post-intervention (week 12), Follow-up (week 24)
  Wearable sensor data features will be extracted from the data such as active and sedentary time, gait speed, and others.

CONTACTS AND LOCATIONS:
Locations (1):
- Rutgers University, Newark, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Yes
Following the completion of this study, the deidentified data set resulting from this body of work will be added to an open source data bank for use by future researchers.
Supporting Information: Analytic Code
Time Frame: The data will become available after study completion. Data availability will be indefinite as it will be posted on a data repository.